CLINICAL TRIAL: NCT04830462
Title: Impact of LTBI Treatment on Glucose Tolerance and Chronic Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Niklas Lorentsson, MD, Herlev and Gentofte Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-20028894 or 126496
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Latent Tuberculosis; Diabetes Mellitus, Type 2
Keywords: low-grade inflammation; glucose metabolism; body composition; cytokines; adipokines; biomarkers
MeSH Terms: conditions — Latent Tuberculosis; Diabetes Mellitus, Type 2 | interventions — Rifampin; Isoniazid; Tablets

STUDY DESIGN:
Intervention Model Description: The study consists of two arms with different patient populations. Both arms will receive identical treatment. Arm A will have type 2 diabetes and latent tuberculosis infection (LTBI). Group B will not have any form of diabetes, but LTBI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTBI and DM (Other): Participants with LTBI and DM will be treated with Rifampicin or Isoniazid at the treating physicians discretion
  Interventions: Drug: Rifampicin 300 Mg Oral Capsule; Drug: Isoniazid 300 Mg ORAL TABLET
- LTBI without DM (Other): Participants with LTBI without DM will be treated with Rifampicin or Isoniazid at the treating physicians discretion
  Interventions: Drug: Rifampicin 300 Mg Oral Capsule; Drug: Isoniazid 300 Mg ORAL TABLET

INTERVENTIONS:
Drug: Rifampicin 300 Mg Oral Capsule — Rifampicin 600 mg orally once daily for 4 months
Drug: Isoniazid 300 Mg ORAL TABLET — Isoniazid 300 mg daily for 6 months

SUMMARY:
This study will be investigating the effect of latent tuberculosis infection (LTBI) treatment on glucose tolerance and low-grade inflammation. Almost a century ago, researchers proposed that diabetes (DM) was associated with increased risk of Tuberculosis infection (TB). A more recent systematic review concluded that DM increases the relative risk for TB 3.1 times. Reversely, TB may affect the glycaemic control; TB is in many cases a chronic infection characterised by long term low-grade inflammation and weight loss, and persons with TB are known to be at risk of hyperglycaemia and DM at time of diagnosis. A latent infection with the m.tuberculosis bacteria is "silent" without symptoms.

1,7 billion have LTBI on a global scale. Event though the infected person does not experience symptoms, increased background inflammation has been shown in LTBI patients in previous studies. We also know that an increase in inflammatory markers precedes clinical development of DM, and that subclinical inflammation contributes to insulin resistance. We hypothesise that LTBI contributes to dysregulated glucose metabolism due to increased low-grade inflammation, and that treatment will reduce low-grade inflammation and improve glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the LTBIDM arm:

* 18+ years
* Known DM type 2

Inclusion criteria for LTBI arm

* 18+ years
* LTBI positive
* No diagnosis with or known DM (1 and 2)

Exclusion Criteria (both arms) :

* Previous treatment for TB or LTBI
* Pregnancy
* Type 1 DM
* Known immunosuppression such as: HIV, steroid treatment within 14 days before inclusion, daily NSAID treatment, ongoing chemotherapy, ongoing immunomodulating treatment or splenectomy
* Known contraindication to both study drugs
* Known active liver disease
* Known severe inflammatory or rheumatological diseases with immune activation and need for prolonged systemic treatment such as IBD, RA, Psoriasis and Wegners granulomatosis
* Recent antibiotic treatment (>2 days) or severe infection within 14 days before enrollment
* Known active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
OGTT (oral glucose tolerance test) | Time Frame: 4-6 months (depending on treatment)
  Reduction in plasma glucose area under the curve during OGTT

SECONDARY OUTCOMES:
Changes in insulin production | Time Frame: 4-6 months (depending on treatment)
  Insulin/c-peptid, HOMA-B pre and post treatment
Changes in insulin resistance | Time Frame: 4-6 months (depending on treatment)
  HOMA-IR pre and post treatment
Changes in low-grade inflammatory markers and in adipokines | Time Frame: 4-6 months (depending on treatment)
  A panel of cytokines and adipokines
INF-gamma change | Time Frame: 4-6 months (depending on treatment)
  Changes in IFN-γ levels after incubation with saline solution, TB antigen or phytohemagglutinin A Pre, during and post treatment
Changes in body composition | Time Frame: 4-6 months (depending on treatment)
  Body composition pre and post treatment measured with DEXA-scanning and/or bioimpedance

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev-Gentofte Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Lorentsson HJN, Clausen CR, Faurholt-Jepsen D, Hansen KB, Ritz C, Jensen SG, Rasmussen EM, Jorgensen A, Lillebaek T, Knop F, Ravn P. The impact of an oral glucose load on IFN-gamma-release in persons infected with Mycobacterium tuberculosis. BMC Infect Dis. 2024 Sep 30;24(1):1079. doi: 10.1186/s12879-024-09920-x. PMID 39350021
- [Derived] Lorentsson HJN, Clausen CR, Faurholt-Jepsen D, Hansen KB, Jensen SG, Krogh-Madsen R, Hagelqvist PG, Johansson PI, Vilsboll T, Knop FK, Ravn P. The effect of Mycobacterium tuberculosis treatment on thrombelastography-assessed haemostasis: a prospective cohort study. Thromb J. 2024 Jun 26;22(1):54. doi: 10.1186/s12959-024-00625-4. PMID 38918780